CLINICAL TRIAL: NCT06371781
Title: Examination of the Relationship Between Sfrp-5, Netrin-4 and Resistin Concentrations in Maternal Blood Samples and Weight Gain During Pregnancy
Brief Title: Examination of the Relationship Between Weight Gain During Pregnancy and Sfrp-5, Netrin-4 and Resistin Concentrations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, ilkin seda can caglayan, assistant professor, Cumhuriyet University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Cumhuriyetobgyn; 1919B012108892 (Other Grant/Funding Number: TUBITAK)
Record Dates: First submitted 2024-04-04; First posted 2024-04-17 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Excessive Weight Gain During Pregnancy
Keywords: Sfrp-5; Netrin-4; Resistin; gestational weight gain
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Intervention Model Description: Pregnant women who were given birth at Cumhuriyet University Faculty of Medicine Hospital Gynecology and Obstetrics Clinic between July 1, 2021 and July 1, 2022 and whose pregnancy follow-ups were performed in our hospital will be included in our prospectively designed study. Researchers will divide the study into two main groups. The first group will consist of pregnant women with above-normal weight gain during pregnancy, and the other group will consist of pregnant women with normal weight gain during pregnancy. It is estimated that 46 control and 44 pregnant women with overweight will be reached during this period. In the study, first a form containing demographic data such as age, education, height and weight will be filled out.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serum Netrin-4, Resistin and Sfrp-5 level measurement (Experimental): In this study, 5 ml of whole blood will be collected from the study group into a biochemistry tube and centrifuged, and the levels of Netrin-4, Resistin and Sfrp-5 in the separated serum will be measured with an ELISA kit.
  Interventions: Diagnostic Test: Serum Netrin-4, Resistin and Sfrp-5 level measurement
- diagnosis of the study group (No Intervention): Individuals who gained excessive weight during pregnancy will be diagnosed as a patient group by evaluating their pre- and post-pregnancy height, weight and BMI values. Those with normal height, weight and BMI values before and after pregnancy will be included in the control group.

INTERVENTIONS:
Diagnostic Test: Serum Netrin-4, Resistin and Sfrp-5 level measurement — Measurements of the levels of these molecules in the serum samples of the study group will be done with the ELISA kit.
  Arms: Serum Netrin-4, Resistin and Sfrp-5 level measurement

SUMMARY:
Researchers thought that the molecules Sfrp-5, Resistin and Netrin-4, which will be examine, they may have a significant effect on weight gain during pregnancy. Based on these foundations, researchers expect changes in the levels of these molecules in women who gain excessive weight during pregnancy. In this study, researchers aimed to examine the moderator relationship between the molecules will be examine and weight gain in women who gained weight above the normal limits determined during pregnancy. For this reason, 44 participant who gained excessive weight during pregnancy and 46 pregnant participant who gained normal weight were included in the study. The levels of Netrin-4, Sfrp-5 and Resistin molecules in the blood serum of the individuals in the study group were measured with a Commercial Elisa kit.

DETAILED DESCRIPTION:
In this study, researchers aimed to examine the moderator relationship between molecules such as Netrin-4, Sfrp-5 and Resistin and weight gain in participant with weight gain above the normal limits determined during pregnancy.

Pregnant participants who were given birth at Cumhuriyet University Faculty of Medicine Hospital Gynecology and Obstetrics Clinic between July 1, 2021 and July 1, 2022 and whose pregnancy follow-ups were performed in our hospital were included in this prospectively designed study. This study was divided into two main groups, the first group will consist of pregnant participant with above-normal weight gain during pregnancy (n = 44), and the other group will consist of pregnant participant with normal weight gain during pregnancy (n = 46). In the study, individuals who agreed to participate in the study were first asked to fill out a form containing demographic data such as age, education, pre- and postnatal height, and weight.

To ensure consistency in women's care, these new Institute of Medicine (IOM) 2009 guidelines are based on BMI cutoffs developed by the World Health Organization and adopted by the National Heart, Lung, and Blood Institute. Weight distribution according to BMI ranges: <18.5 kg/m2 (underweight), 18.5-24.9 kg/m2 (normal weight), 25-29.9 kg/m2 (overweight) and ≥30 kg/m2 (obese). According to these guidelines, the recommended weight gain range for underweight (UW) women is 12.5-18 kg, for normal weight (NW) women 11.5-16 kg and overweight women (OW) 7-11.5 kg, obese ( OB) women are recommended to gain only 5-9 kg during pregnancy. These values according to the IOM-2009 guideline are the most widely accepted recommendations for weight gain during pregnancy. Weight gain above these values researchers have specified will be considered as excessive weight gain for us.The levels of these molecules in the serum of the study groups were measured using a commercial ELISA kit.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnant women over 37 weeks
* Without metabolic disorders
* Do not use medication
* Healthy fetuses and mom

Exclusion Criteria:

* pregestational diabetes,
* gestational diabetes
* hypertension and related metabolic diseases
* twin pregnancies,
* pregnancies under 37 weeks
* with large babies

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Obtaining blood serum for measurement of serum Sfrp-5, Netrin-4 and Resistin | one day
  Blood will be taken from individuals only once; therefore, minor redness and swelling may occur at the site where blood is taken; other than that, there is no serious risk. The measured molecules will be measured in blood serum and there will be no intervention other than blood collection from individuals.Measurements of these three molecules will be measured simultaneously in a single blood sample.

SECONDARY OUTCOMES:
Calculating BMI (kg/m^2) from height (m) and weight (kg) measurement values for diagnosis. | one day
  Pre-pregnancy height (m) and weight (kg) measurements of pregnant women participating in the study will be learned and these values will be used to calculate pre-pregnancy BMI. Height (m) and weight (kg) values will be measured as soon as they are included in the study and will be used to calculate pregnancy BMI. There is no risk to individuals.

CONTACTS AND LOCATIONS:
Overall Officials: İlkin Seda CAN ÇAĞLAYAN, Asso.Prof., Study Director — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No